CLINICAL TRIAL: NCT01252771
Title: Phosphate Kinetic Modeling 2
Acronym: PKM2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fresenius Medical Care North America (Industry)
Collaborators: Renal Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-188
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2011-06

CONDITIONS: Hyperphosphatemia; ESRD
Keywords: phosphorus; dialysis; PhosLo
MeSH Terms: conditions — Hyperphosphatemia; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PKM report and algorithm (Experimental): Phosphate kinetic modeling was performed and displayed in graphical form laboratory results and an estimated phophorus protein ratio
  Interventions: Other: PKM Algorithm

INTERVENTIONS:
Other: PKM Algorithm — The subject's serum calcium and phosphorus values will be input into PKM in order to determine the required PhosLo prescription. The prescription is determined as the number of gelcaps per day that must be taken by the subject.
  If PKM determines the number of PhosLo gelcaps per day to be greater than or equal to the subject's current prescription, then PKM will calculate the current Ca++ and phosphate balance. Furthermore, the PKM algorithm will determine the additional number of PhosLo gelcaps needed to achieve neutral phosphate (P) balance with serum P reduced to 5.5 mg/dL.
  The PKM algorithm also calculates the total P intake between dialyses and along with ePCR also calculates a Phosphorus/Protein Ratio (PPR). This ratio ranges from 8 to 14 in dialysis patients following a renal diet.

SUMMARY:
The study aims to investigate the concept of computer based Phosphate Kinetic Modeling (PKM) in the hemodialysis patient population. This computerized algorithm model was developed as a tool to aid physicians in controlling a hemodialysis patient's phosphate level. Once a subject consents to participate in the study, the subject's dietary phosphate intake will be estimated by the modeling program and the appropriate dose of the phosphate binder calcium acetate (PhosLo) will be recommended accordingly. If necessary, the Ca++ concentration of the dialysate will be changed to remove any excess calcium absorbed as the result of an increase in the PhosLo prescription to control phosphorus.

DETAILED DESCRIPTION:
PKM consists of a set of validated and computerized algorithms to perform the following steps:

1. Calculate calcium (Ca) and phosphorus (P) intake and absorption in individual patients as a function of the prescribed doses of Vitamin D analogues, protein catabolic rate (PCR) and dietary and binder Ca intakes.
2. Calculate P removal between dialyses by P binders and P and Ca removal during dialysis from kinetic analysis of total P and Ca transport during dialysis based on dialyzer P and Ca transport coefficients and the levels of dialysate Ca and serum Ca and P.
3. Thus from analysis of intake, absorption and removal the program can calculate net Ca and P balance in modeled patients.
4. Calculate the daily dose of phosphate binder (PhosLo) required to reduce the serum P to normal in patients with hyperphosphatemia.
5. Calculate the dialysate Ca required to achieve zero calcium balance over complete dialysis cycles - the interdialytic interval and immediately succeeding dialytic interval.
6. The program also computes a Phosphorus-Protein ratio (PPR, the total P removed divided by PCR, mg/gm/day) which provides a quantitative index of compliance with prescribed dietary P restriction and/or the prescribed dose of binders. It is hoped that this information will be valuable to guide semi-quantitative evaluations of diet P and binder intakes in patients difficult to manage. Study subjects will bring their PhosLo pill bottles to treatments weekly. At this time the subject's dietitian will determine and record the remaining pills. The comparison of pills taken versus pilled prescribed will be performed with any data available. While weekly counts are desirable for providing more information about the consistency of a patient's compliance, a minimum of monthly counts will be sufficient. This will be done to validate the PPR range needed to accurately identify compliance with PhosLo regimen. Patients will also be instructed to bring all empty PhosLo bottles to site dietitian. The site dietitian will record pill count data in a form for each patient. The updated version of the PKM algorithm also includes computation of the dose of vitamin D analogues and cinacalcet (Sensipar). This modification of the PKM algorithm may help to better achieve neutral calcium balance, because the intestinal calcium absorption heavily depends on vitamin D levels. The computation of cinacalcet aids the control of parathyroid hormone (PTH) levels within the target range.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is capable of giving informed consent.
2. Age > 18 years
3. Thrice weekly hemodialysis with a dialysate Ca++ concentration (CdiCa) of 2.0, 2.25 or 2.5 mEq/L
4. Stable CdiCa of either 2.0, 2.25 or 2.5 mEq/L for ≥ 4 weeks
5. Dialysis vintage ≥ 3 months
6. Three-month average P > 5.5 mg/dL AND 2 of 3 monthly average P >=5.8 mg/dL
7. Patients currently prescribed calcium acetate (PhosLo) mono-therapy , sevelamer monotherapy, or a combination therapy of PhosLo plus sevelamer for phosphate binding with willingness of physician to switch to PhosLo monotherapy
8. Fresenius Optiflux F 160, 180 or 200 dialyzer

Exclusion Criteria:

1. Any laboratory abnormality, medical condition or psychiatric disorder which in the opinion of the investigator would put the subject's disease management at risk or may result in the subject being unable to comply with study requirements
2. Known pregnancy
3. Parathyroidectomy
4. iPTH < 50 pg/mL
5. Hospitalization in past 30 days
6. Dialysate potassium prescription other than 2 or 3 mmol/L
7. Serum Ca++ < 7.5 mg/dL
8. Current vitamin D therapy using calcitriol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
change in serum phosphorus | 6 months
  The primary outcome variable is the change in serum phosphorus between a baseline period and the latest value of the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kotanko, MD, Principal Investigator — Renal Research Institute
Locations (1):
- Renal Research Insitutue, New York, New York, United States